CLINICAL TRIAL: NCT04299412
Title: Diagnostic Accuracy of the DPP Fever Panel II Asia and the DPP Micro Reader
Brief Title: Diagnostic Accuracy of the DPP II Assay
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: FE005
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Febrile Illness; Melioidosis; Diagnoses Disease
MeSH Terms: conditions — Melioidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Melioidosis cases: serum samples collected from patients with B. pseudomallei positive cultures
  Interventions: Device: DPP Fever Panel II assay
- Non-melioidosis cases: serum samples collected from patients with B. pseudomallei negative cultures
  Interventions: Device: DPP Fever Panel II assay

INTERVENTIONS:
Device: DPP Fever Panel II assay — Multiplex lateral flow immunoassay (DPP® Fever Panel II Assay) that is able to detect (i) antigens produced by Dengue, Zika, Chikungunya, Malaria and Burkholderia and (ii) IgM directed against Dengue, Zika, Chikungunya, Leptospira, Rickettsia typhi and Orientia tsutsugamushi. The assay comes with a reader that provides results interpretation to the operator in a few seconds

SUMMARY:
Burkholderia pseudomallei is responsible for melioidosis, a disease that can present a range of signs and symptoms and can be treated by a specific drug regimen. Diagnosis of melioidosis is made by isolation of the bacteria from body fluids or tissues such as blood, skin or sputum. Although this is considered the gold standard, bacterial isolation has low diagnostic sensitivity, requires specific infrastructures (biosafety level 3 laboratories) and skilled staff that are not always available in LMICs. This may lead to inappropriate patient management and care.

Chembio, in partnership with FIND, has developed a multiplex lateral flow immunoassay (DPP® Fever Panel II Assay) that is able to detect antigens from common causes of febrile illnesses, included Burkholderia. FIND will conduct a laboratory study in Menzies Health School of Research to estimate the diagnostic accuracy of the DPP II Assay using retrospective samples that are positive for B. pseudomallei. Results will help in estimating the diagnostic accuracy of the assay for this pathogen.

ELIGIBILITY:
Inclusion Criteria:

- Samples that can be included in the trial must have been collected exclusively during the "Assessment of a New Rapid Diagnostic Test for Melioidosis" study (HREC 04/09) conducted by the Menzies School of Health Research. They must be well-characterized with confirmation of presence or absence of B. pseudomallei by bacterial culture.

Exclusion Criteria:

* Samples with volume <120 µL
* Samples collected during projects other than the HREC 04/09 project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sera samples were collected between December 2014 and June 2018 for the "Assessment of a New Rapid Diagnostic Test for Melioidosis" study that was conducted by the Menzies School of Health Research in Darwin, Australia. Patients recruited during that study presented to the Royal Darwin Hospital (RDH) with suspicion of melioidosis and consented to provide blood samples and to allow their use in diagnostic studies. Their samples are stored at -80°C in the Tropical and Emerging Infectious Diseases laboratory at the Menzies School of Health Research.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity, with 95% confidence intervals, for the detection of B. pseudomallei by the DPP assay in comparison to a reference standard. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Menzies School of Health Research, Darwin, Australia

IPD SHARING:
Plan to Share IPD: Undecided